CLINICAL TRIAL: NCT03267459
Title: Prediction of the Response Using Dynamic Contrast-enhanced Magnetic Resonance Imaging Before Intra-arterial Chemotherapy in Children With Retinoblastoma
Brief Title: Can Pretreatment MRI be Used to Predict Intra-arterial Chemotherapy Response in Retinoblastoma?
Acronym: PREDIR
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2017_2
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dynamic contrast-enhanced MRI — Dynamic contrast-enhanced perfusion sequences added to MRI examination performed at the beginning of intra arterial chemotherapy.

SUMMARY:
Retinoblastoma is the most frequent intraocular tumor in children and represents 6% of all pediatric cancers before the age of 5 years-old. The outcome is now excellent with 95 to 97% of 5-years survival rate. Conservative treatments are being more and more used, and intra arterial chemotherapy is one of the adjuvant treatments proposed to the children. The treatment is efficient in most cases, but a small proportion of children will have an early progression after treatment. MRI is used for the diagnosis of retinoblastoma. We aim to find prognostic factors using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) for early identification of children response to intra arterial chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* grade B to D retinoblastoma
* prescription of intra arterial chemotherapy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with retinoblastoma, undergoing intra arterial chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
response to chemotherapy | 18 months
  Persistence of ocular scarring (= favorable outcome)18 months after the end of the treatment by intra-arterial chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Augustin Lecler, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation A De Rothschild, Paris, France